CLINICAL TRIAL: NCT03950531
Title: The Effect of Bronchiectasis on the Exacerbation and Mortality of Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Bronchiectasis on the Exacerbation and Mortality in COPD
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, Zeynep FENDOGLU, Principal investigator, Ministry of Health, Turkey
Other Study IDs: 123678
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Bronchiectasis; Chronic Obstructive Pulmonary Disease
Keywords: Bronchiectasis; Chronic Obstructive Pulmonary Disease; Exacerbation; Computed Tomography
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD exacerbation without Bronchiectasis: COPD patients who have been in exacerbation period and have no bronchiectasis
  Interventions: Other: No intervention
- COPD exacerbation with Bronchiectasis: COPD patients who have been in exacerbation period and have bronchiectasis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease of the airways and lungs that develops against harmful particles or gases with exacerbations. Coexistence of bronchiectasis with COPD may lead to worsening of the functional parameters as well as alteration of the microbiological pattern in exacerbations and may negatively affect the exacerbation result parameters.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease of the airways and lungs that develops against harmful particles or gases with exacerbations. COPD exacerbations are characterized by worsening of dyspnea, coughing and expectoration. Exacerbations requiring hospitalization are the main cause of morbidity and mortality in COPD. Bronchiectasis is the irreversible extension of the bronchi. Usually follows with chronic sputum cough, airway obstruction and recurrent infection episodes. The association of bronchiectasis and COPD has long been known and its incidence is in the range of 30-50%. Coexistence of bronchiectasis with COPD may lead to worsening of the functional parameters as well as alteration of the microbiological pattern in exacerbations and may negatively affect the exacerbation result parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent thoracic tomography in the last year according to index exacerbation date were included in the study

Exclusion Criteria:

* Cases that mimic COPD exacerbation (pneumonia, pulmonary thromboembolism, pulmonary congestion, pneumothorax, pleural effusion, lung malignancy, asthma, asthma-COPD overlap syndrome) and patients admitted to the intensive care unit were excluded from the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COPD exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-01-25 (Actual); Primary Completion 2014-12-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Charlson Comorbidity Index | 1 hour
  Comorbidity scores

SECONDARY OUTCOMES:
Spirometry | 1 hour
  Pulmonary function measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Kokturk, Professor, Study Chair — Gazi University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No